CLINICAL TRIAL: NCT02750787
Title: An Evaluation of the Use of a Peptide-based Formula in an Adult Population
Brief Title: Use of a Peptide-based Formula in an Adult Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DA12
Record Dates: First submitted 2016-04-19; First posted 2016-04-26 (Estimated); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Malabsorption
MeSH Terms: conditions — Malabsorption Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nutritional Study Product (Experimental): A ready-to-drink peptide-based liquid formula for patients with impaired gastro-intestinal function.
  Interventions: Other: Nutritional Study Product

INTERVENTIONS:
Other: Nutritional Study Product — Two 220 ml servings per day

SUMMARY:
The study is designed to observe the use of a peptide-based oral nutrition supplement in adults with chronic malabsorption or maldigestion who require supplemental nutrition as assessed by a clinician.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age.
* Subject has chronic malabsorption or maldigestion.
* Subject requires supplemental nutrition as assessed by a clinician.
* Subject agrees to consume 2 servings of the study product a day for at least 16 consecutive days during Treatment period.

Exclusion Criteria:

* Subject is currently taking or has taken antibiotics within 2 weeks prior to enrollment in the study.
* Subject has current active malignant disease or was treated within the last 6 months for cancer.
* Subject has a history of diabetes mellitus.
* Subject is pregnant as demonstrated by a urine pregnancy test.
* Subject has severe auto immune disease and is on immuno-modulating therapy.
* Subject has a history of allergy to any of the ingredients in the study product.
* Subject has active HIV.
* Subject has a known aversion to flavor of product being tested.
* Subject has known dementia, brain metastases, eating disorders, history of significant neurological or psychiatric disorder, or any other psychological condition that may interfere with study product consumption.
* Subject has an obstruction of the gastrointestinal tract precluding ingestion or absorption of the study product.
* Subject is taking part in another non-Sponsor approved clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Study Product Consumption | Day 1 to Day 23
  Subject Diary

SECONDARY OUTCOMES:
Body Mass Index | Change from Screening to Day 23
  Calculated from Height and Weight
Medication Use | Screening to Study Day 23
  Subject Interview of Dose, Unit and Frequency
Adverse Events | Screening to Day 25

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Nelson, PhD, Study Chair — Abbott Nutrition
Locations (1):
- St. Boniface Hospital, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Undecided